CLINICAL TRIAL: NCT00370565
Title: Efficacy And Safety Of Exubera (Inhaled Insulin) Therapy In Subjects With Type 2 Diabetes Mellitus Not Well Controlled With Combination Oral Agents: A Three-Month, Outpatient, Parallel Comparative Trial.
Brief Title: Effect on Glycemic Control of Inhaled Insulin Alone or Added to Dual Oral Therapy After Failure of Dual Oral Therapy.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: Sanofi (Industry); Nektar Therapeutics (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 217-109
Record Dates: First submitted 2006-08-29; First posted 2006-08-31 (Estimated); Last update posted 2007-02-13 (Estimated); Status verified 2007-02

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

INTERVENTIONS:
Drug: Inhaled Human Insulin

SUMMARY:
To assess the impact on glucose control by inhaled insulin alone or added to two oral anti-diabetic agents in patients with type 2 diabetes who are not well controlled on 2 oral anti-diabetic agents.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 Diabetes Mellitus as defined by American Diabetes Association (ADA) at least 1 year earlier.
* Patients were required to have been treated with a stable oral agent regimen involving 2 antidiabetc medications: 1 insulin secretagogue (a sulfonylurea or replabinide) and 1 insulin sensitizer (a thiazolidinedione or metformin).

Exclusion Criteria:

* Asthma, COPD
* Smoking during the previous 6 months

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 345
Dates: Start 1999-06; Study Completion 2000-09

PRIMARY OUTCOMES:
The primary efficacy endpoint is the change from baseline HbA1c measured at 12 weeks after randomization.
HbA1c is measured at Weeks -4, -1, 0, 6, and 12 of comparative treatment. The baseline value is the mean of the Week -1 and Week 0 values.

SECONDARY OUTCOMES:
Secondary: Efficacy: change in fasting plasma glucose and meal glucose response (2-h postprandial increment in plasma glucose)Fasting plasma glucose measured at Weeks -4, -1, 0, and 12 (the Weeks -1 and 12 measurements will be part of the meal studies)
Meal glucose response measured at Week -1 and at Week 12;
These results for efficacy are measured in the lab using plasma samples collected during clinic visits,
not the subject's home glucose monitoring results.
Comparison of 24-hour home glucose profiles.
Proportion of subjects with acceptable or good glycemic control (e.g., HbA1c < 8.0% or <7.0%) at the end of treatment, incidence and severity of hypoglycemic episodes, discontinuation rate, change in fasting lipid profile, and change in body weight.
A patient satisfaction and preference questionnaire will be administered at screening, at baseline, during active therapy, and at the end of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (41):
- United States (32):
  - Pfizer Investigational Site, Irvine, California
  - Pfizer Investigational Site, Long Beach, California
  - Pfizer Investigational Site, Los Angeles, California
  - Pfizer Investigational Site, Newport Beach, California
  - Pfizer Investigational Site, San Diego, California
  - Pfizer Investigational Site, Tustin, California
  - Pfizer Investigational Site, New Britain, Connecticut
  - Pfizer Investigational Site, New Haven, Connecticut
  - Pfizer Investigational Site, Washington D.C., District of Columbia
  - Pfizer Investigational Site, Clearwater, Florida
  - Pfizer Investigational Site, Hollywood, Florida
  - Pfizer Investigational Site, Miami, Florida
  - Pfizer Investigational Site, Tampa, Florida
  - Pfizer Investigational Site, Louisville, Kentucky
  - Pfizer Investigational Site, New Orleans, Louisiana
  - Pfizer Investigational Site, Minneapolis, Minnesota
  - Pfizer Investigational Site, Columbia, Missouri
  - Pfizer Investigational Site, St Louis, Missouri
  - Pfizer Investigational Site, Omaha, Nebraska
  - Pfizer Investigational Site, New York, New York
  - Pfizer Investigational Site, Rochester, New York
  - Pfizer Investigational Site, Greenville, North Carolina
  - Pfizer Investigational Site, Winston-Salem, North Carolina
  - Pfizer Investigational Site, Cleveland, Ohio
  - Pfizer Investigational Site, Portland, Oregon
  - Pfizer Investigational Site, Philadelphia, Pennsylvania
  - Pfizer Investigational Site, Austin, Texas
  - Pfizer Investigational Site, Dallas, Texas
  - Pfizer Investigational Site, Irving, Texas
  - Pfizer Investigational Site, San Antonio, Texas
  - Pfizer Investigational Site, Burlington, Vermont
  - Pfizer Investigational Site, Renton, Washington
- Canada (9):
  - Pfizer Investigational Site, Calgary, Alberta
  - Pfizer Investigational Site, Edmonton, Alberta
  - Pfizer Investigational Site, Red Deer, Alberta
  - Pfizer Investigational Site, Winnipeg, Manitoba
  - Pfizer Investigational Site, St. John's, Newfoundland and Labrador
  - Pfizer Investigational Site, Halifax, Nova Scotia
  - Pfizer Investigational Site, Ottawa, Ontario
  - Pfizer Investigational Site, Toronto, Ontario
  - Pfizer Investigational Site, Laval, Quebec

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=109&StudyName=Effect+on+Glycemic+Control+of+Inhaled+Insulin+Alone+or+Added+to+Dual+Oral+Therapy+after+Failure+of+Dual+Oral+Therapy%2E